CLINICAL TRIAL: NCT05973461
Title: Effects of Exercise With Virtual Reality on Females and Males With or Without Depression
Brief Title: Effects of Exercise and Virtual Reality on Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: analyzing data
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Judy Wilson, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-0376
Record Dates: First submitted 2023-05-11; First posted 2023-08-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Symptoms of Depression
MeSH Terms: conditions — Depression | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: males and females, with and without symptoms of depression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cycle Ergometer and Virtual Reality (Experimental): 30 min ride on cycle ergometer while viewing neighborhood scenes using virtual reality
  Interventions: Device: Exercise and virtual reality
- Cycle Ergometer (Experimental): 30 min ride on cycle ergometer
  Interventions: Other: Riding a cycle ergometer

INTERVENTIONS:
Device: Exercise and virtual reality — Riding a cycle ergometer while experiencing virtual reality
  Arms: Cycle Ergometer and Virtual Reality
Other: Riding a cycle ergometer — Riding on a cycle ergometer without experiencing virtual reality
  Arms: Cycle Ergometer

SUMMARY:
This study is evaluating the effects of riding on a cycle ergometer while experiencing virtual reality to determine its effect on mood.

DETAILED DESCRIPTION:
Adults (males and females) above the age of 18 yrs will be recruited to determine if they have symptoms of depression based on a questionnaire (Center for Epidemiologic Studies - Depression Scale (CES-D). They will then complete a Beck Inventory before and after the exercise. Participants will be divided into groups either having symptoms of depression or not. They will be randomized to ride on a cycle ergometer with or without using Virtual Reality (VR) that will allow them to view neighborhoods or parks during the exercise. The ergometer will be set at resistance raising the heart rate to 65% of their age-predicted heart rate maximum. They will ride for 20 min and then complete the Beck Inventory to determine any changes in their depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years
* With or without symptoms of depression
* Physically inactive or sedentary (less than 30 minutes per day)
* Normal vision and no color blindness
* No physical disorders such as walking with assistance

Exclusion Criteria:

* Below the age of 18 years or over 65 years,
* Women who are pregnant
* Individuals who have been diagnosed with mental disorders
* Individuals with leg injuries
* Individuals with cardiac problems
* Individuals with a history of asthma
* Individuals with a body mass index over 30.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory Scale of Measurement | 5 minutes
  Assessment of symptoms of depression pre and post-intervention cycle exercise. The Beck Depression Inventory is a 21-item, multiple-choice, self-report survey that measures characteristic attitudes and symptoms of depression. The score range is 0-63. The higher the score the more severe the depression. Scores above 41 are considered "extreme depression."
Spatial Working Memory (SWM) | 8 minutes
  A measure of the key aspects of working memory and storage of information over short periods of time.
Neuropsychological Outcomes: Motor Screen Tasks (MOT) | 3 minutes
  MOT provides a general indication that psychomotor function is intact enough to proceed with more sophisticated cognitive testing:

SECONDARY OUTCOMES:
Neuropsychological Outcomes: MOT Mean Latency, MOT Total Correct, and MOT Total Errors | 10 minutes
  This test is a general assessment of whether there are sensorimotor deficits or lack of comprehension. Outcome is measured by reaction time in milliseconds of the participant reaching out and touching the "X" correctly (in the middle of the X) on the tablet in response to the stimulus. The maximum score is 6000 milliseconds. The number of total correct touches and total errors in not touching correctly out of 10 are recorded. Ex: MOT mean latency = 927.9 ml +/- 131.43 ms; MOT Total Correct = 10; MOT Total Errors = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Judy R Wilson, Ph.D., Principal Investigator — UTArlington
Locations (1):
- UTArlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No